CLINICAL TRIAL: NCT07185893
Title: A Multicenter, Open-label, Randomized Controlled Trial Evaluating the Efficacy and Safety of Romiplostim N01 in the Treatment of Thrombocytopenia Associated With Concurrent/Sequential Chemoradiotherapy and Chemotherapy Combined With/Without Immunotherapy in Solid Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jun wang (Other)
Responsible Party: Sponsor-Investigator, Jun wang, Director of radiotherapy department1, Hebei Medical University Fourth Hospital
Organization: Hebei Medical University Fourth Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025KY020
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor Malignancies, Cancer; CTIT-Chemotherapy Induced Thrombocytopenia; Thrombocytopenia
Keywords: Romiplostim N01; Human Interleukin-11; solid tumor; thrombocytopenia; CTIT
MeSH Terms: conditions — Neoplasms; Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Romiplostim N01 (Experimental): Administer Romiplostim N01 subcutaneously in the abdominal area. The initial dose is 3 μg/kg, once a week. The subsequent dose will be adjusted according to the patient's platelet count
  Interventions: Drug: Romiplostim N01
- Human Interleukin-11 (Active Comparator): Human Interleukin-11 for Injection (rhlL-11) 25 - 50 μg/kg, subcutaneous injection, once a day, for at least 7 - 10 days.
  Interventions: Drug: Human Interleukin-11

INTERVENTIONS:
Drug: Human Interleukin-11 — Human Interleukin-11 for Injection (rhlL-11) 25 - 50 μg/kg, subcutaneous injection, once a day, for at least 7 - 10 days.
  Arms: Human Interleukin-11
Drug: Romiplostim N01 — Administer Romiplostim N01 subcutaneously in the abdominal area. The initial dose is 3 μg/kg, once a week. The subsequent dose will be adjusted according to the patient's platelet count
  Arms: Romiplostim N01

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and efficacy of Romiplostim N01 in patients with solid tumors who are undergoing concurrent/sequential radiotherapy and chemotherapy（combined with/without immunotherapy）-related thrombocytopenia.

All eligible patients will be stratified and randomly assigned based on baseline platelet count（Stratification factors: whether the baseline platelet count of the patients is greater than 50×10^9/L. ） . All patients will be randomly assigned in a 1:1 ratio to experimental group or control group:

Experimental group: Romiplostim N01 (N=53) Control group：Human Interleukin-11(rhlL-11) (N=53) The main questions this trial aims to answer are: 1. The proportion of patients who received platelet transfusion due to thrombocytopenia during the treatment process, as well as the adjustment, delay and discontinuation of radiotherapy and chemotherapy doses； 2. Can patients treated with Romiplostim N01 restore their platelet count to ≥ 100×10^9/L and what is the response rate of patients during the treatment (response criteria: no need for platelet transfusion and PLT increase ≥ 50×10^9/L or at least twice the baseline or PLT increase to ≥ 100×10^9/L)；3. The safety and tolerance of Romiplostim N01 in treating CTIT.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 to 80 years old (man or female);
2. Confirmed with solid tumor by pathological histology or cytology examination;
3. The patient is undergoing concurrent/sequential radiotherapy ± immunotherapy;
4. During the treatment period, the patient experienced a decrease in platelets, and the platelet count within the last 3 days before enrollment was 25×10^9/L < platelet count ≤ 75×10^9/L;
5. The estimated survival period at screening is ≥ 3 months, and it is expected that the current chemotherapy cycle can be used for ≥ 2 cycles;
6. ECOG 0 - 2;
7. Fully understand and comply with the requirements of this study, and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Platelet count ≤ 25×10^9/L at baseline;
2. The patient has previously received treatments for thrombocytopenia, such as thrombopoietin receptor agonists (TOP-RA), recombinant human thrombopoietin (rhTPO), or rhIL-11, etc.;
3. Patients with hematological disorders, including lymphoma, leukemia, aplastic anemia, primary immune thrombocytopenia, myelodysplastic syndromes, multiple myeloma, and myelodysplastic syndrome, etc.;
4. Have experienced thrombocytopenia due to non-tumor treatment within the past 6 months, including but not limited to EDTA-dependent pseudo-thrombocytopenia, splenomegaly, infection, bleeding, etc.;
5. After red blood cell or erythropoietin (EPO) infusion, hemoglobin is still < 50g/L, or after granulocyte colony-stimulating factor (G-CSF) treatment, absolute neutrophil count is still < 1.0×10^9/L;
6. Have experienced any arterial or venous thrombosis within the past 6 months;
7. Have suffered from severe cardiovascular diseases (such as NYHA cardiac function class III-IV), increased risk of thrombosis-related arrhythmias (such as atrial fibrillation), coronary artery stent implantation, angioplasty, and coronary artery bypass grafting within the past 6 months;
8. Have received platelet transfusion within 5 days before randomization or enrollment;
9. Patients with positive hepatitis C antibody and excessive HCV-RNA detection, positive hepatitis B surface antigen and excessive HBV-DNA detection, patients with severe cirrhosis, positive HIV antibody, or positive syphilis antibody;
10. During screening, for subjects without liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are ≥ 3 times ULN; for subjects with liver metastasis, ≥ 5 times ULN;
11. Serum creatinine concentration ≥ 1.5 times ULN or eGFR ≤ 60ml/min;
12. Patients who are allergic or intolerant to the active ingredient or excipients of Romiplostim N01 for injection;
13. Planning to get pregnant or in the lactation period;
14. The investigator determines that the patient is not suitable to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieved a response within 14 days of treatment | The assessment will be conducted 31 months after the start of the treatment.
  Response criteria: no need for platelet transfusion and PLT increase ≥ 50×10^9/L or at least twice the baseline level or PLT increase to ≥ 100×10^9/L.

SECONDARY OUTCOMES:
The median time for platelet count to recover to ≥ 100 × 10^9/L | The assessment will be conducted 31 months after the start of the treatment.
The proportion of patients who received platelet transfusions during the treatment stage due to thrombocytopenia | The assessment will be conducted 31 months after the start of the treatment.
The proportion of patients who achieved a response within 3 days, 7 days, and 10 days of treatment | The assessment will be conducted 31 months after the start of the treatment.
  Response criteria: no need for platelet transfusion and PLT increase ≥ 50×10^9/L or at least twice the baseline level or PLT increase to ≥ 100×10^9/L.
The incidence of dose adjustment, delay, or termination of radiotherapy and chemotherapy due to thrombocytopenia | The assessment will be conducted 31 months after the start of the treatment.
Incidence rate of adverse events | The assessment will be conducted 40 months after the start of the treatment.
  The adverse events of the Romiplostim N01 and Human Interleukin-11 will be evaluated, Including the incidence of all adverse events, grade 3/4 adverse events, the incidence of adverse events leading to treatment discontinuation, leading to death, SAEs, as well as the duration of adverse events, management measures and outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No